CLINICAL TRIAL: NCT03092869
Title: Effects of Feet and Ankle Mobilization on Balance of Older Adults
Acronym: FEET_BALANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Hernández, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DHG01
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Aging Problems
Keywords: Feet; Ankle; Balance; Manual Therapy; Older Adult

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Feet and Ankle Mobilization
  Interventions: Other: Feet and Ankle Mobilization; Other: Proprioceptive Training
- Control Group (Active Comparator): Proprioceptive Training
  Interventions: Other: Proprioceptive Training

INTERVENTIONS:
Other: Feet and Ankle Mobilization — A set of manual therapy mobilization in feet and ankle joints
  Arms: Experimental Group
Other: Proprioceptive Training — A set of proprioceptive exercises oriented to improve balance abilities

SUMMARY:
This study aims to assess whether mobilization of the ankle and foot produces significant improvements in the balance of the elderly.

To this end, a randomized study was designed with a control group that performs proprioception exercises and an experimental group that also performs a mobilization of the ankle and foot joints.

DETAILED DESCRIPTION:
Aging leads to a decrease in physical activity and a reduction of postural control, which implies a loss of balance control, both static and dynamic, thus compromising the autonomy of the elderly and increasing the risk of suffering a fall. It has been observed that the balance degenerates in an accelerated way from 60 years of age. Basically appears a natural physiological degeneration of the organism, which affects strength, range of mobility, reduces vestibular function, there is loss vision and lower cardiopulmonary capacity.

In the older adult who suffers falls, in relation to the one who does not suffer, a series of differences or determinants have been observed. In this group, a series of characteristics such as the lower flexibility of the ankle joint and the muscle-tendon complex are present, hallux valgus appears, lower foot tenderness or a decrease in the strength in the first plantar flexor finger. They appear to have poorer balance and have less force in the flexors of the soles accompanied by less mobility of the foot inversion-eversion.

One of the causes that seems to contribute in the decrease of the balance in the older adult are the alterations in the ankle and foot, besides supposing a worse capacity of adaptation to the possible environmental changes. Before a deficit of this type, the subject tends to compensate for his position with compensatory strategies in other joints of the lower limb. It has also been shown that as we grow older, there is an increase in the demand for articulation of the other joints, such as the hip and knee, secondary to a decrease in joint range of ankle and foot or weakness of the dorsal flexors of the foot.

It follows that there is a relationship between alterations in the ankle and foot and the balance in the elderly, all related to the forces that suffer the ankle in the gait and to the low normal activity. Any alteration in this joint could predetermine an alteration of its function in maintaining stability in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Old adults over 60 years

Exclusion Criteria:

* Subjects with balance disorders whether vestibular or central.
* Subjects with lower limb prosthesis.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-09-02 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | Change from baseline to end of intervention (one month)
  This is a 14 item scale used to assess the overall state of balance of the oder adult

SECONDARY OUTCOMES:
Test Up and Go | Change from baseline to end of intervention (one month)
  It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Pressure Platform Outcome | Change from baseline to end of intervention (one month)
  Romberg test. Static balance when standing in the platform in a static position without moving the feet during 30 seconds
Range of Movement | Change from baseline to end of intervention (one month)
  Flexion-extension range of movement of the ankle joint

CONTACTS AND LOCATIONS:
Overall Officials: David Hernández, PT, Principal Investigator — University of Valencia
Locations (2):
- Spain (2):
  - Universidad de Valencia, Valencia
  - University of Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided